CLINICAL TRIAL: NCT03939741
Title: Evaluation of Therapeutic Potential of Stromal Vascular Fraction (Autologous Adipose Derived Mesenchymal Stem Cell) Based Treatment for Chronic Kidney Disease
Brief Title: SVF (Adipose Tissue Derived MSC) Based Therapy for CKD.
Acronym: StemCell&CKD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangladesh Laser & Cell Surgery Institute & Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BangladeshLCS001
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic kidney disease; Stromal vascular fraction; Adipose derived stem cell
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Participants will be placed in a single group. Those having a harvested total "Adipose Derived Stem Cell (ADSC)" count (in 5 ml SVF solution) above 1 x 10^6 will be included in the study and they will be studied for Phase I/ Phase II trial by the proposed outcome measures over the stipulated time frame.
  Those having a harvested total "Adipose Derived Stem Cell (ADSC)" count (in 5 ml SVF solution) less than 1 x 10^6 will be excluded from the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Participants having a harvested total "Adipose Derived Stem Cell (ADSC)" count (in 5 ml SVF solution) more than 1 x 10^6.
  Genetic: SVF containing Autologous Non Expanded ADSC.
  Interventions: Biological: SVF Containg Autologous Non Expanded ADSC

INTERVENTIONS:
Biological: SVF Containg Autologous Non Expanded ADSC — 5 ml of SVF containing Autologous Non Expanded ADSC will be injected intravenously and outcome will be observed over the period of 1(one) year.

SUMMARY:
1. To assess the safety of stromal vascular fraction (Autologous Non-Expanded ADSC) injection in patients with Chronic Kidney Disease (CKD).
2. To assess the efficacy of stromal vascular fraction (Autologous Non-Expanded ADSC) injection in patients with Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
Introduction:

Chronic kidney disease (CKD) is a disease of alarmingly increasing prevalence (8 - 16%) associated with mortality [1]. CKD can progress towards end-stage renal disease (ESRD), requiring renal replacement therapy. ESRD currently accounts for 6.3% of Medicare spending in the United States and is projected to increase by 85% by 2015 [2]. In a study conducted among the rural populations in Bangladesh overall CKD prevalence was found about 19% [3]. Furthermore, ESRD has a major impact on quality of life and life expectancy [4]. Therefore, it is very important to develop therapeutic interventions to prevent, alleviate, or decelerate the progression of renal failure.

Diabetes mellitus and hypertension represent major causes of CKD and initiation of dialysis [5]. In addition, glomerular diseases, malnutrition, infectious diseases, and acute kidney injury may lead to ESRD, contributing to the increased global burden of death [6]. Current treatment modalities often fail to target the major underlying contributors to the progression of renal disease [7]. Management of CKD at present mostly aims at control of the predisposing factors and supplementation of kidney homeostatic functions but not at the treatment of the diseased kidney itself. Again due to lack of adequate facilities or financial constraints people of a developing country like Bangladesh are unable to continue long-term or lifelong dialysis. Chronic glomerular and tubule-interstitial fibrosis is a common pathway to ESRD, often associated with apoptosis, oxidative damage, fibrosis, and microvascular rarefaction. Unfortunately, the regenerative potential of kidneys is limited under chronic conditions and inefficient to prevent progressive glomerulosclerosis and tubule-interstitial fibrosis [8]. Treatment strategies that boost cellular regeneration might therefore offer good alternatives for patients with CKD.

Stromal vascular fraction (SVF):

SVF of adipose tissue is a rich source of pre-adipocytes, mesenchymal stem cells (MSC), endothelial progenitor cells, T cells, B cells, mast cells as well as adipose tissue macrophages [9,10]. SVF is a component of the lipo-aspirate obtained from liposuction of subcutaneous tissue. Lipo-aspirate contains a large population of stem cells called adipose-derived stem cells (ADSCs), which share a number of similarities with bone marrow stem cells, including the capacity for multilineage differentiation.

Stem Cells:

A stem cell is a generic term referring to any unspecialized cell that is capable of long-term self-renewal through cell division but that can be induced to differentiate into a specialized, functional cell. Stem cells are generally two types, embryonic stem cells, and adult stem cells. Adult stem cells can be obtained from many differentiated tissues including bone marrow, bone, fat, muscle etc. Obtaining adult stem cells also does not raise any ethical concerns [11]. For most studies, the adult stem cell in question is actually a mesenchymal stem cell (MSC) or mesenchymal stromal cell. They are multipotent but not pluripotent, which means they can differentiate into some, or "multiple," but not all tissue types [11]. Stem cells that are harvested from the patient with the intention of administering them back to the same patient are termed autologous MSCs. MSC can also be isolated from the bone marrow (bmMSC), peripheral blood, connective tissue, skeletal muscle, the dental pulp (dpMSC), umbilical cord wall (ucMSC), umbilical cord blood (cbMSC), amniotic fluid (afMSC) and all have been used in experimental settings to treat various types of renal diseases. An important feature of MSCs is their capacity to induce the proliferation of renal glomerular and tubular cells, increasing cellular survival [12].

Advantages of adipose tissue-derived stem cells (ADSCs):

ADSCs are somatic stem cell populations contained in fat tissue and have been shown to possess stem cell properties such as trans-differentiation and self-renewal [13]. Similar to other types of MSCs, ADSCs express multiple CD marker antigens (CD73+CD90+CD105+ CD34+/- CD11b- CD104b- CD19- CD31- CD45- SMA-) [14,15]. Additionally, utilizing ADSCs is advantageous in that large quantities of stem cells are easily isolated using minimally invasive surgical procedures [16].

ADSCs are vascular precursor cells. Many studies have shown that SVF contains progenitor cells that are able to differentiate into endothelial cells and participate in blood vessel formation [17]. Additionally, a recent study demonstrated that SVF cells expressing both pericyte and mesenchymal markers reside in a peri-endothelial location and stabilize endothelial networks [17] Another study showed that ADSCs were transplanted into an ischemic renal cortex preferentially migrate toward microvessels where they differentiate into vascular smooth muscle cells [18]. Some trials on kidney transplant recipients as well as the one on FSGS and 2 on CKD patients include in their protocol the utilization of adMSC. Adipose tissue is an important source of MSC, with a frequency 100 to 1000 times higher than bmMSC. They also seem to possess a higher potential for angiogenesis or vasculogenesis [19].

Kidney disease and mesenchymal stem cells:

A number of different types of cells from the bone marrow have been tested in animals and in clinical studies for potential use in kidney disease. Amongst all the cells under investigation, MSCs have shown the most promising results to date as they help kidney cells to grow, inhibit cell death, and encourage the kidney's own stem cells to repair kidney damage [20].

Few clinical trials have tested the safety and efficacy of MSCs for renal disease. Reinders and colleagues studied safety and feasibility in six kidney allograft recipients who received two intravenous infusions of expanded autologous bone marrow-derived MSCs [21]. Importantly, delivery of autologous MSCs was not associated with adverse events, nor did it compromise graft survival. Several clinical trials are currently underway to evaluate the therapeutic potential of autologous and allogeneic MSCs for the treatment of renal diseases [22] Administration of both bmMSC and adMSC has demonstrated significant renoprotective effects including reduction of intrarenal inflammatory infiltrate, decreased fibrosis, and glomerulosclerosis [12] MSCs possess unique immunomodulatory properties that ameliorate inflammation and immune responses, constituting a promising tool to facilitate renal repair. In recent years, experimental studies have uncovered the potential of MSCs to improve renal function in several models of CKD, and several clinical studies have indicated their safety and efficacy in CKD [22].

ADSCs could be incorporated into damaged tissues or organs which could give rise to new functional components and also exert potent anti-inflammatory, anti-fibrotic, or immunomodulation effects through paracrine or autocrine routes (via vascular endothelial growth factor, granulocyte/macrophage colony-stimulating factor, stromal-derived factor-1alpha, and hepatocyte growth factor) [23,24]. Interestingly, it is proposed that even apoptotic or dying ADSCs exhibit distinctive immunosuppressive properties [25]. ADSCs have been shown to possess stronger anti-inflammatory and immuno-modulating functions than bone marrow-derived MSCs [26].

Villanueva et al. explored the effect of ADSCs on CKD by a single intravenous infusion of ADSCs on a nephrectomy-induced CKD model of rats [27]. ADSC treatment was associated with reduced plasma creatinine, higher levels of epitheliogenic and angiogenic proteins, and improved renal function. Work by Hyun et al [28] illustrated the beneficial effects of ADSCs on improving renal function in an IgAN mouse model. Zhang et al. [30] found that repeated systemic administration of ADSCs attenuated proteinuria, glomerulus hypertrophy, and tubular interstitial injury in a DN rat model [29].

Currently, several clinical trials have been uploaded to the NIH database, all aiming to test mainly the safety of using MSC and their efficacy in treating CKD. Two of them propose the use of autologous bmMSC and two adMSC. A study conducted in Tehran, the Islamic Republic of Iran, was designed to provide confirmation of Mesenchymal stem cell therapy in CKD. There 18 months of safety and efficacy of autologous MSC as a therapy for CKD total of 10 patients were conducted with I/V injection of a high dose of 2x106/kg of autologous MSC. Assessments were performed at 1,3,6,12 and 18 months after cell injections [30].

Another study was conducted in Birmingham, Alabama, Rochester, Minnesota, and Jackson, Mississippi, the USA where a stem cell product called "Mesenchymal stem cell" grown from a person's own fat tissue was infused back into the patient's own kidney and primary outcome measured after 3 months where renal tissue oxygenation increased and decrease in kidney inflammation was seen as a secondary outcome [31].

Route of delivery:

Various routes for delivery of ADSCs, ADSC-induced cells, or ADSCs combined with compound materials have been developed for the treatment of different diseases or damaged tissue. These routes can be classified into two categories: systemic delivery through blood vessels (intravenous injection or intra-arterial injection) or local delivery directly into injured tissues or organs [32] The route of MSC delivery may influence the cells' capacity to home and engraft the damaged tissue, and thereby their efficacy for renal repair. Commonly used experimental methods to deliver MSCs include systemic intravenous, intra-arterial, or intra-parenchymal delivery. In nonhuman primates, the cells distribute broadly into the kidneys, skin, lung, thymus, and liver with estimated levels of engraftment ranging from 0.1 to 2.7% [33].

The route of MSC delivery, intravenous, intra-arterial, or intra-parenchymal, may affect their efficiency for kidney repair. When labeled MSC intravenously infused into baboons were observed for 9-21 months, estimated levels of engraftment in the kidney, lung, liver, thymus, and skin ranged from 0.1-2.7% [34] Indeed, the intravenous route lags in delivery efficiency, because MSC may initially be trapped in the lungs. Intra-arterial infusion of MSC was the most effective route to achieve immunomodulation in rat kidney transplantation, possibly by avoiding lodging in the pulmonary circulation, allowing MSC to home to the injured kidney [35].

An important feature of MSCs is their capacity to induce the proliferation of renal glomerular and tubular cells, increasing cellular survival. By secreting proangiogenic and trophic factors, injected MSCs not only can enhance proliferation but also can decrease the apoptosis of tubular cells [36]. Several routes of administration (intra-parenchymal, sub-capsular, intravenous) have been explored and all seem to be effective. Multiple, repeated injections of MSCs appear to be even more effective than single injections [37,38].

Methodology:

A Prospective study from April 2019 onwards (Approximately Five years or till completion of sample requirements with a minimum of one year of follow-up) will be conducted in Bangladesh LASER & Cell Surgery Institute & Hospital, Dhaka. Thirty-One patients with CKD who fulfill the selection criteria and are admitted to the selected health care facility for treatment will be included in the study. SVF (stromal vascular fraction) will be collected from the abdominal subcutaneous adipose tissue. Subsequent processing ( Incubation, centrifugation, mixing, washing & neutralization ) will produce the final viable & active SVF (ADSCs) cell which will be transfused intravenously. Considering the possibility of further damage to the already damaging or damaged kidney during angiography and placement of a catheter into the renal artery, the investigators opt for intravenous transfusion of the SVF. Before transfusion samples will be collected & cell counting will be done using an automated fluorescent cell counter.

ELIGIBILITY:
Inclusion Criteria:

* A patient is eligible for the study if all of the followings apply:

  1. Aged 18-80 years (inclusive)
  2. With chronic kidney disease (CKD)stage 3 to 5 (eGFR 60 to 0 mL/min/1.73m2 (inclusive)) Note : eGFR = estimated glomerular filtration rate
  3. Having provided informed written consent.

Exclusion Criteria:

Any patient meeting any of the exclusion criteria will be excluded from study participation.

1. Known hypersensitivity to any component used in the study.
2. With inadequate hematologic function with: absolute neutrophil count (ANC) <1,500/μL OR platelets < 100,000/μL OR Hemoglobin < 8 g/dL
3. With impaired hepatic function with: serum bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase (AKP), prothrombin time above and normal reference and serum albumin below normal reference range.
4. With hemoglobin A1c (HbA1c) > 8.0%
5. With serious prior or ongoing medical conditions (e.g. concomitant illness such as cardiovascular (e.g. New York Heart Association grade III or IV), hepatic e.g. Child-Pugh Class C), psychiatric condition, alcoholism, drug abuse), medical history, physical findings, ECG findings, or laboratory abnormality that in the investigators' opinion could interfere with the results of the trial or adversely effect the safety of the patient
6. Pregnant or lactating women or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period
7. With known history of human immunodeficiency virus (HIV) infection or any type of hepatitis
8. Judged to be not applicable to this study by investigator such as difficulty of follow-up observation
9. With any other serious diseases/medical history considered by the investigator not in the condition to enter the trial
10. Known or suspected abuse of alcohol or narcotics
11. With known history of cancer within past 5 years
12. With any autoimmune disease
13. With congenital kidney disease
14. With precancerous condition or with raised tumour markers like Alpha feto protein, Carcino embryonic antigen (CEA), C.A 19.9, C.A 125, Serum PSA above normal reference range.
15. Parcipants having a harvested total "Adipose Derived Stem Cell (ADSC)" count (in 5 ml SVF solution) less than 1 x 10^6 will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of minor adverse events (MAEs) , serious adverse events (SAEs) which may be immediate, early or late - for Phase I | Week 48
  Minor adverse events (MAEs):
  1. Pain from lipo-suction > 7 days (Early)
  2. Fever > 7 days (Early)
  3. Subcutaneous hematoma / abscess formation (Early)
  4. Allergic reaction (Immediate)
  Serious adverse events (SAEs)
  1. Anaphylaxis (Immediate)
  2. Pulmonary embolism or infarction (Immediate)
  3. Outset of any neoplastic change (Late)
  4. Outset of new Cardiovascular events (Late)
  5. Outset of new Cerebrovascular or neurological events (Late)
  6. Reactivation of treated tuberculosis (Late)
Change from baseline to 24 week visit in glomerular filtration rate (GFR) and split renal function in all patients - for Phase II | Weeks 0, 24
  GFR with split renal function will be evaluated using DTPA Renogram.
Change from baseline to 24 week visit in estimated glomerular filtration rate (eGFR) with serum creatinine level in patients with CKD 4 and below - for Phase II | Weeks 0, 2, 4, 12, 24
  eGFR will be calculated by Serum Creatinine level using MRDR formula during all visits.
Change from baseline to 24 week visit in need for dialysis in patients with CKD 5 - for phase II | Weeks 0, 2, 4, 12, 24
  Need for dialysis is described as
  1. No dialysis needed - Score 0
  2. Randomly (more than 6 days interval) - Score 1
  3. At 6 (six) days interval / Once weekly - Score 2
  4. At 5 (five) days interval - Score 3
  5. At 4 (four) days interval - Score 4
  6. At 3 (three) days interval / 2 times a week - Score 5
  7. At 2 (two) days interval - Score 6
  8. At 1 (one) day interval / every alternate day./ 3 times a week - Score 7

SECONDARY OUTCOMES:
Change from baseline to all post-treatment visits in body weight | Weeks 0, 2, 4, 12, 24, 36, 48
  Weight in Kg will be recorded for each patient during each follow up
Change from baseline to all post-treatment visits in Blood-pressure | Weeks 0, 2, 4, 12, 24, 36, 48
  Blood pressure will be measured in each patient during each follow up
Change from baseline to all post-treatment visits in S.creatinine | Weeks 0, 2, 4, 12, 24, 36, 48
  1. S. Creatinine level will be measured during each follow up.
  2. In case of patients having dialysis Pre and Post dialysis S. Creatinine levels will be measured at or near follow up dates.
Change from baseline to all post-treatment visits in blood urea. | Weeks 0, 2, 4, 12, 24, 36, 48
  Blood Urea will be measured in all patients during each follow up.
Change from baseline to all post-treatment visits in Hemoglobin level | Weeks 0, 2, 4, 12, 24, 36, 48
  1. Hemoglobin level will be measured in gm/dl and percentage
  2. Need for blood transfusion will be recorded
  3. Need for erythropoietin will be recorded
Change from baseline to all post-treatment visits in urine microalbumin-to-creatinine ratio (UMCR) | Weeks 0, 2, 4, 12, 24, 36, 48
  Urinary Microalbumin and creatinine will be measured in each patient during each follow up
Change from baseline to all post-treatment visits in hemoglobin A1c | Weeks 0, 2, 4, 12, 24, 36, 48
  HbA1C will be measured in each patient during each follow up
Change from baseline to all post-treatment visits in random blood sugar (RBS) | Weeks 0, 2, 4, 12, 24, 36, 48
  RBS will be measured in each patient during each follow up
Change from baseline to all post-treatment visits in Anti-Hypertensive medication if there is any. | Weeks 0, 2, 4, 12, 24, 36, 48
  All anti hypertensive medicines with their doses will be recorded including any changes in each patient during each follow up
Change from baseline to all post-treatment visits in Hypoglycemic agent if there is any. | Weeks 0, 2, 4, 12, 24, 36, 48
  All hypoglycemic agents including their doses with any changes will be recorded for all diabetic patients during each follow up
Change from baseline to post-treatment visits in urine total protein-creatinine ratio (UPCR) | Weeks 0, 24, 48
  Urinary total protein and Creatinine ratio will be done in each patient during each follow up
Change from baseline to all post-treatment visits in urinary Protein-to-creatinine ratio PCR) | Weeks 0, 2, 4, 12, 24, 36, 48
  Urinary Protein and creatinine will be measured in each patient during each follow up
Change from baseline to post-treatment level of serum Alpha Feto Protein | Weeks 0, 24, 48
  Serum Alpha Feto protein will be measured as a tumour marker for Hepato-cellular carcinoma and also Tumour of Testis and Ovary.
Change from baseline to post-treatment level of serum CEA level | Weeks 0, 24, 48
  Serum CEA level will be measured as a tumour marker for Colo-rectal Carcinoma and also for Cancer of Stomach, pancreas, breast, lungs, thyroid and ovary.
Change from baseline to post-treatment level of serum CA 19.9 level | Weeks 0, 24, 48
  Serum C.A 19.9 level will be measured as a tumour marker for Pancreatic Carcinoma
Change from baseline to post-treatment level LDH level | Weeks 0, 24, 48
  Serum LDH level will be measured as tumour marker for Lymphoma
Change from baseline to post-treatment level of Beta 2 Microglobulin level | Weeks 0, 24,48
  Serum Beta 2 Microglobulin level will be measured as a prognostic tool, as CKD patients invariably has a raised serum level.
Change from baseline to post-treatment level of serum CA 125 level (in case of female patients) | Weeks 0, 24, 48
  Serum C.A 125 level will be measured as a tumour marker for Ovarian Cancer
Change from baseline to post-treatment level of PSA level (in case of male patients) | Weeks 0, 24,48
  Serum PSA level will be measured as a tumour marker for Prostatic Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Md. Firoj Khan, MBBS,FRCP,MD, Principal Investigator — Bangladesh Laser and Cell Surgery Institute and Hospital, Dhaka, Bangladesh.; Dr. Mohammed Yakub Ali MBBS, MPhil, MSc, PhD, Study Chair — Bangladesh Laser and Cell Surgery Institute and Hospital, Dhaka, Bangladesh.; Dr. Jahangir Md. Sarwar, MBBS, FCPS, Study Director — Bangladesh Laser and Cell Surgery Institute and Hospital, Dhaka, Bangladesh.
Locations (1):
- Bangladesh Laser And Cell Surgery Institute And Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] Gilbertson DT, Liu J, Xue JL, Louis TA, Solid CA, Ebben JP, Collins AJ. Projecting the number of patients with end-stage renal disease in the United States to the year 2015. J Am Soc Nephrol. 2005 Dec;16(12):3736-41. doi: 10.1681/ASN.2005010112. Epub 2005 Nov 2. PMID 16267160
- [Background] Prevalence of Chronic Kidney Disease (CKD) and Identification of Associated risk Factors among Rulral Population by Mass Screening. Hasan MJ , Kashem MA,, Rahman MH, Quddhush R , Rahman M, Sharmeen A, Islam N. CBMJ 2012;1(1):20-26.
- [Background] Wyld M, Morton RL, Hayen A, Howard K, Webster AC. A systematic review and meta-analysis of utility-based quality of life in chronic kidney disease treatments. PLoS Med. 2012;9(9):e1001307. doi: 10.1371/journal.pmed.1001307. Epub 2012 Sep 11. PMID 22984353
- [Background] Collins AJ, Foley RN, Chavers B, Gilbertson D, Herzog C, Johansen K, Kasiske B, Kutner N, Liu J, St Peter W, Guo H, Gustafson S, Heubner B, Lamb K, Li S, Li S, Peng Y, Qiu Y, Roberts T, Skeans M, Snyder J, Solid C, Thompson B, Wang C, Weinhandl E, Zaun D, Arko C, Chen SC, Daniels F, Ebben J, Frazier E, Hanzlik C, Johnson R, Sheets D, Wang X, Forrest B, Constantini E, Everson S, Eggers P, Agodoa L. 'United States Renal Data System 2011 Annual Data Report: Atlas of chronic kidney disease & end-stage renal disease in the United States. Am J Kidney Dis. 2012 Jan;59(1 Suppl 1):A7, e1-420. doi: 10.1053/j.ajkd.2011.11.015. No abstract available. PMID 22177944
- [Background] Perico N, Remuzzi G. Chronic kidney disease: a research and public health priority. Nephrol Dial Transplant. 2012 Oct;27 Suppl 3:iii19-26. doi: 10.1093/ndt/gfs284. Epub 2012 Jul 3. No abstract available. PMID 22764188
- [Background] Rivera JA, O'Hare AM, Harper GM. Update on the management of chronic kidney disease. Am Fam Physician. 2012 Oct 15;86(8):749-54. PMID 23062158
- [Background] Benigni A, Morigi M, Remuzzi G. Kidney regeneration. Lancet. 2010 Apr 10;375(9722):1310-7. doi: 10.1016/S0140-6736(10)60237-1. PMID 20382327
- [Background] Riordan NH, Ichim TE, Min WP, Wang H, Solano F, Lara F, Alfaro M, Rodriguez JP, Harman RJ, Patel AN, Murphy MP, Lee RR, Minev B. Non-expanded adipose stromal vascular fraction cell therapy for multiple sclerosis. J Transl Med. 2009 Apr 24;7:29. doi: 10.1186/1479-5876-7-29. PMID 19393041
- [Background] Schipper HS, Prakken B, Kalkhoven E, Boes M. Adipose tissue-resident immune cells: key players in immunometabolism. Trends Endocrinol Metab. 2012 Aug;23(8):407-15. doi: 10.1016/j.tem.2012.05.011. Epub 2012 Jul 12. PMID 22795937
- [Background] Reinders ME, Fibbe WE, Rabelink TJ. Multipotent mesenchymal stromal cell therapy in renal disease and kidney transplantation. Nephrol Dial Transplant. 2010 Jan;25(1):17-24. doi: 10.1093/ndt/gfp552. Epub 2009 Oct 26. PMID 19861311
- [Background] Peired AJ, Sisti A, Romagnani P. Mesenchymal Stem Cell-Based Therapy for Kidney Disease: A Review of Clinical Evidence. Stem Cells Int. 2016;2016:4798639. doi: 10.1155/2016/4798639. Epub 2016 Sep 19. PMID 27721835
- [Background] Kokai LE, Rubin JP, Marra KG. The potential of adipose-derived adult stem cells as a source of neuronal progenitor cells. Plast Reconstr Surg. 2005 Oct;116(5):1453-60. doi: 10.1097/01.prs.0000182570.62814.e3. PMID 16217495
- [Background] Lin CS, Xin ZC, Deng CH, Ning H, Lin G, Lue TF. Defining adipose tissue-derived stem cells in tissue and in culture. Histol Histopathol. 2010 Jun;25(6):807-15. doi: 10.14670/HH-25.807. PMID 20376787
- [Background] Lin F. Adipose tissue-derived mesenchymal stem cells: a fat chance of curing kidney disease? Kidney Int. 2012 Oct;82(7):731-3. doi: 10.1038/ki.2012.158. PMID 22975993
- [Background] Huixi Li1, 2, Guiting Lin1*, and Tom F Lue1 Potential application of adipose tissue-derived stem cells for urological disease. Bladder 2014;1(1). DOI: 10.14440/bladder.2014.23
- [Background] Stashower M, Smith K, Williams J, Skelton H. Stromal progenitor cells present within liposuction and reduction abdominoplasty fat for autologous transfer to aged skin. Dermatol Surg. 1999 Dec;25(12):945-9. doi: 10.1046/j.1524-4725.1999.99098.x. PMID 10594628
- [Background] Halvorsen YC, Wilkison WO, Gimble JM. Adipose-derived stromal cells--their utility and potential in bone formation. Int J Obes Relat Metab Disord. 2000 Nov;24 Suppl 4:S41-4. doi: 10.1038/sj.ijo.0801503. PMID 11126240
- [Background] Moseley TA, Zhu M, Hedrick MH. Adipose-derived stem and progenitor cells as fillers in plastic and reconstructive surgery. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):121S-128S. doi: 10.1097/01.prs.0000234609.74811.2e. PMID 16936551
- [Background] Kidney disease: how could stem cells help?. http://www.eurostemcell.org /factsheet/kidney-disease-how-could-stem-cells-help
- [Background] Reinders ME, de Fijter JW, Roelofs H, Bajema IM, de Vries DK, Schaapherder AF, Claas FH, van Miert PP, Roelen DL, van Kooten C, Fibbe WE, Rabelink TJ. Autologous bone marrow-derived mesenchymal stromal cells for the treatment of allograft rejection after renal transplantation: results of a phase I study. Stem Cells Transl Med. 2013 Feb;2(2):107-11. doi: 10.5966/sctm.2012-0114. Epub 2013 Jan 24. PMID 23349326
- [Background] Eirin A, Lerman LO. Mesenchymal stem cell treatment for chronic renal failure. Stem Cell Res Ther. 2014 Jul 4;5(4):83. doi: 10.1186/scrt472. PMID 25158205
- [Background] Rehman J, Traktuev D, Li J, Merfeld-Clauss S, Temm-Grove CJ, Bovenkerk JE, Pell CL, Johnstone BH, Considine RV, March KL. Secretion of angiogenic and antiapoptotic factors by human adipose stromal cells. Circulation. 2004 Mar 16;109(10):1292-8. doi: 10.1161/01.CIR.0000121425.42966.F1. Epub 2004 Mar 1. PMID 14993122
- [Background] Meliga E, Strem BM, Duckers HJ, Serruys PW. Adipose-derived cells. Cell Transplant. 2007;16(9):963-70. doi: 10.3727/096368907783338190. PMID 18293895
- [Background] Thum T, Bauersachs J, Poole-Wilson PA, Volk HD, Anker SD. The dying stem cell hypothesis: immune modulation as a novel mechanism for progenitor cell therapy in cardiac muscle. J Am Coll Cardiol. 2005 Nov 15;46(10):1799-802. doi: 10.1016/j.jacc.2005.07.053. Epub 2005 Oct 17. PMID 16286162
- [Background] Banas A, Teratani T, Yamamoto Y, Tokuhara M, Takeshita F, Osaki M, Kawamata M, Kato T, Okochi H, Ochiya T. IFATS collection: in vivo therapeutic potential of human adipose tissue mesenchymal stem cells after transplantation into mice with liver injury. Stem Cells. 2008 Oct;26(10):2705-12. doi: 10.1634/stemcells.2008-0034. Epub 2008 Jun 5. PMID 18535155
- [Background] Villanueva S, Carreno JE, Salazar L, Vergara C, Strodthoff R, Fajre F, Cespedes C, Saez PJ, Irarrazabal C, Bartolucci J, Figueroa F, Vio CP. Human mesenchymal stem cells derived from adipose tissue reduce functional and tissue damage in a rat model of chronic renal failure. Clin Sci (Lond). 2013 Aug;125(4):199-210. doi: 10.1042/CS20120644. PMID 23480877
- [Background] Quimby JM, Webb TL, Habenicht LM, Dow SW. Safety and efficacy of intravenous infusion of allogeneic cryopreserved mesenchymal stem cells for treatment of chronic kidney disease in cats: results of three sequential pilot studies. Stem Cell Res Ther. 2013 Apr 30;4(2):48. doi: 10.1186/scrt198. PMID 23632128
- [Background] Zhang L, Li K, Liu X, Li D, Luo C, Fu B, Cui S, Zhu F, Zhao RC, Chen X. Repeated systemic administration of human adipose-derived stem cells attenuates overt diabetic nephropathy in rats. Stem Cells Dev. 2013 Dec 1;22(23):3074-86. doi: 10.1089/scd.2013.0142. Epub 2013 Aug 21. PMID 23844841
- [Background] Papazova DA, Oosterhuis NR, Gremmels H, van Koppen A, Joles JA, Verhaar MC. Cell-based therapies for experimental chronic kidney disease: a systematic review and meta-analysis. Dis Model Mech. 2015 Mar;8(3):281-93. doi: 10.1242/dmm.017699. Epub 2015 Jan 29. PMID 25633980
- [Background] Malaga-Dieguez L, Bouhassira D, Gipson D, Trachtman H. Novel therapies for FSGS: preclinical and clinical studies. Adv Chronic Kidney Dis. 2015 Mar;22(2):e1-6. doi: 10.1053/j.ackd.2014.10.001. PMID 25704355
- [Background] You D, Jang MJ, Lee J, Suh N, Jeong IG, Sohn DW, Kim SW, Ahn TY, Kim CS. Comparative analysis of periprostatic implantation and intracavernosal injection of human adipose tissue-derived stem cells for erectile function recovery in a rat model of cavernous nerve injury. Prostate. 2013 Feb 15;73(3):278-86. doi: 10.1002/pros.22567. Epub 2012 Jul 20. PMID 22821215
- [Background] Ezquer FE, Ezquer ME, Parrau DB, Carpio D, Yanez AJ, Conget PA. Systemic administration of multipotent mesenchymal stromal cells reverts hyperglycemia and prevents nephropathy in type 1 diabetic mice. Biol Blood Marrow Transplant. 2008 Jun;14(6):631-40. doi: 10.1016/j.bbmt.2008.01.006. Epub 2008 Apr 14. PMID 18489988
- [Background] Fischer UM, Harting MT, Jimenez F, Monzon-Posadas WO, Xue H, Savitz SI, Laine GA, Cox CS Jr. Pulmonary passage is a major obstacle for intravenous stem cell delivery: the pulmonary first-pass effect. Stem Cells Dev. 2009 Jun;18(5):683-92. doi: 10.1089/scd.2008.0253. PMID 19099374
- [Background] Zonta S, De Martino M, Bedino G, Piotti G, Rampino T, Gregorini M, Frassoni F, Dal Canton A, Dionigi P, Alessiani M. Which is the most suitable and effective route of administration for mesenchymal stem cell-based immunomodulation therapy in experimental kidney transplantation: endovenous or arterial? Transplant Proc. 2010 May;42(4):1336-40. doi: 10.1016/j.transproceed.2010.03.081. PMID 20534295
- [Background] Bi B, Schmitt R, Israilova M, Nishio H, Cantley LG. Stromal cells protect against acute tubular injury via an endocrine effect. J Am Soc Nephrol. 2007 Sep;18(9):2486-96. doi: 10.1681/ASN.2007020140. Epub 2007 Jul 26. PMID 17656474
- [Background] Lee SR, Lee SH, Moon JY, Park JY, Lee D, Lim SJ, Jeong KH, Park JK, Lee TW, Ihm CG. Repeated administration of bone marrow-derived mesenchymal stem cells improved the protective effects on a remnant kidney model. Ren Fail. 2010;32(7):840-8. doi: 10.3109/0886022X.2010.494803. PMID 20662698
- [Background] Semedo P, Correa-Costa M, Antonio Cenedeze M, Maria Avancini Costa Malheiros D, Antonia dos Reis M, Shimizu MH, Seguro AC, Pacheco-Silva A, Saraiva Camara NO. Mesenchymal stem cells attenuate renal fibrosis through immune modulation and remodeling properties in a rat remnant kidney model. Stem Cells. 2009 Dec;27(12):3063-73. doi: 10.1002/stem.214. PMID 19750536

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT03939741/Prot_SAP_ICF_001.pdf